CLINICAL TRIAL: NCT03897946
Title: Evaluating Immunogenicity of a Birth Dose of HBV Vaccine in the DRC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The American Society of Tropical Medicine and Hygiene (Other); Burroughs Wellcome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-2793
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants and care providers will not be masked, but the investigators and data analysts will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Hepatitis B exposed, with birth dose (Experimental): The 100 HBV-exposed (born to HBsAg-positive mothers) infants who are already enrolled in the parent AVERT study will also be enrolled in the current study, as the "HBV-exposed cohort" (Group A). These exposed infants will not receive additional interventions on top of the AVERT study since they will already be receiving a birth dose vaccine through the AVERT study.
  Interventions: Biological: Birth dose hepatitis B vaccine
- Group B: Hepatitis B unexposed, no birth dose (No Intervention): For the "HBV-unexposed cohort" in this study, the investigators will enroll 200 infants born to HBsAg-negative mothers. Half (100) of these infants will receive the routine three-dose series of HBV vaccine according to the standard EPI schedule in the DRC with no additional birth dose vaccine (Group B).
- Group C: Hepatitis B unexposed, with birth dose (Experimental): Group C will consist of the other half (100) of infants in the "HBV-unexposed cohort" who will receive four doses of HBV vaccine including a birth dose vaccine prior to the routine EPI schedule.
  Interventions: Biological: Birth dose hepatitis B vaccine

INTERVENTIONS:
Biological: Birth dose hepatitis B vaccine — Groups A and C will receive a birth dose of hepatitis B vaccine within 24 hours of life.
  Arms: Group A: Hepatitis B exposed, with birth dose; Group C: Hepatitis B unexposed, with birth dose

SUMMARY:
This project will assess the immunogenicity of a birth dose of hepatitis B vaccine in hepatitis B-exposed and hepatitis B-unexposed infants in Kinshasa, Democratic Republic of the Congo. A better understanding of the protection offered by the addition of birth dose vaccine to the EPI schedule is necessary in order to promote universal adoption of a birth dose vaccine in the DRC and throughout SSA.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) remains a neglected tropical disease despite the availability of effective prevention measures. HBV vaccine has been incorporated into pediatric immunization schedules worldwide for nearly two decades, and yet 257 million people are still living with chronic HBV infection. Current control measures are failing to prevent further transmission of HBV, especially in sub-Saharan Africa (SSA), where hepatitis B surface antigen (HBsAg) prevalence surpasses 8% in highly endemic areas. An estimated 1% of infants (>365,000 per year) are infected with HBV by mother-to-child transmission (MTCT) in SSA, and when infected in the first year of life, these infants have a 90% risk of developing chronic infection.

Pediatric HBV is a substantial problem in the Democratic Republic of the Congo (DRC). Preliminary data from the 2013-2014 Demographic and Health Survey in the DRC revealed that 2.2% of children under the age of five are infected with HBV.

Why is the seroprevalence of HBV so high in children? The three-dose HBV vaccine has been part of the Expanded Program on Immunization (EPI) in the DRC since 2007, with vaccination rates now approaching 80%. However, the EPI vaccination schedule does not begin until six weeks of life. In contrast, in developed countries, infants receive the first dose of HBV vaccine at birth. This birth dose is rarely administered in SSA. Routine birth dose vaccination could be a simple and cost-effective means to reduce the pool of infected and highly infectious children in the DRC.

While the protective efficacy of a three-dose series of HBV vaccine plus immunoglobulin (HBIG) initiated at birth is ≥95%, immunogenicity of HBV vaccine administered according to the EPI schedule (pentavalent vaccine administered at 6,10 and 14 weeks) is only 80-85%. This gap in antibody response leads to a significant population of children who are potentially vulnerable to infection in infancy or later in life. The immunogenicity of a four-dose HBV vaccine series including a monovalent birth dose prior to the EPI schedule has not been fully assessed to date. Furthermore, HBIG is not available in SSA due to prohibitive cost and storage issues, necessitating an evaluation of the effectiveness of the vaccine series alone without HBIG.

In collaboration with the DRC Ministry of Health, Abbott Laboratories and Ohio State University, the investigators are conducting the Arresting Vertical Transmission of HBV (AVERT-HBV) study, which leverages the existing HIV PMTCT framework in the DRC to screen and treat pregnant women and their infants to prevent MTCT of HBV. The investigators will use the AVERT study population to recruit participants (HBV-exposed infants and their mothers) for this study. Women who screen negative for HBV as part of AVERT will be included in this study as the HBV-unexposed cohort.

While HIV PMTCT programs have been successful in reducing the number of HIV-infected infants in the DRC, many infants fall into the HIV-exposed uninfected (HEU) category. These HEU infants are known to have lowered immune responses to vaccines than HIV-unexposed infants, including protective immunity to HBV after the EPI-associated three-dose series. Little is known about the effects of in utero HBV exposure on the immune response to HBV vaccine. The investigators hypothesize that because the immune response of infants exposed to HBV may be blunted, these infants may benefit from an additional dose of HBV vaccine at birth.

Using the AVERT-HBV cohort as a basis, this project will assess the immunogenicity of the birth dose vaccine in HBV-exposed and HBV-unexposed infants. A better understanding of the protection offered by the addition of birth dose vaccine to the EPI schedule is necessary in order to promote universal adoption of a birth dose vaccine in the DRC and throughout SSA.

This prospective cohort study will involve 100 HBV-exposed infants who will receive 4 doses of HBV vaccine starting at birth (Group A), 100 HBV-unexposed infants who receive 3 doses of HBV vaccine according to the EPI schedule (Group B) and 100 HBV-unexposed infants who receive 4 doses of HBV vaccine starting at birth (Group C). The infants will be followed for 12 months, at which time protective immunity against HBV, defined as HBsAb ≥10 milli-international units (mIU)/mL, will be measured.

ELIGIBILITY:
MOTHERS

Inclusion Criteria

* HBsAg+ mothers and HBsAg- mothers will be recruited from the cohort screened during the AVERT study at 2 maternity centers (Binza and Kingasani) in Kinshasa.

Exclusion Criteria

* Any women who do not intend to stay in Kinshasa for prenatal care through delivery or who deliver at a facility other than Binza or Kingasani
* Women <18 years of age

INFANTS

Inclusion Criteria

* Infants born to HBsAg-positive and HBsAg-negative women who receive care at Binza and Kingasani maternity centers will be recruited for participation in this study.

Exclusion Criteria

* HIV-exposed infants (those born to HIV-positive mothers) will be excluded given an expected difference in immune response in these infants and inability to recruit enough HIV-exposed infants to be able to detect these differences in immune response
* HBV-unexposed infants weighing <2,000 grams at birth will not be eligible to receive the birth HBV vaccine. (HBV-exposed infants receive the birth dose vaccine regardless of birth weight because the potential benefit of preventing mother-to-child transmission outweighs the potential risk of vaccination in a low birthweight infant. The research team recognizes that Group B may include a disproportionate number of low birthweight infants compared to Group C, but will account for this in post-hoc analyses and if need be, will exclude low birthweight infants from the analysis to account for potential bias).
* Infants born at a facility other than one of the two maternity centers

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 569 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Proportion of Infants with Protective Immunity | At 12 months of age
  Protective immunity is defined as quantitative HBsAb ≥ 10 milli-International unit(mIU)/mL

SECONDARY OUTCOMES:
Proportion of Infants with Adverse Reactions to the Birth Dose Hepatitis B Vaccine | Within 2-3 days after birth
  Adverse reactions will include fever, fatigue and injection site soreness, as described in the Package Insert (https://www.fda.gov/downloads/biologicsbloodvaccines/vaccines/approvedproducts/ucm224503.pdf). Infants will be monitored for adverse reactions for safety purposes during the time they spend with their mothers at the maternity center after birth (expected average stay of 2-3 days).

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Meshnick, MD, PhD, Study Director — UNC-Chapel Hill; Peyton J Thompson, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Binza and Kingasani Maternity Centers, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Hara GA, McNaughton AL, Maponga T, Jooste P, Ocama P, Chilengi R, Mokaya J, Liyayi MI, Wachira T, Gikungi DM, Burbridge L, O'Donnell D, Akiror CS, Sloan D, Torimiro J, Yindom LM, Walton R, Andersson M, Marsh K, Newton R, Matthews PC. Hepatitis B virus infection as a neglected tropical disease. PLoS Negl Trop Dis. 2017 Oct 5;11(10):e0005842. doi: 10.1371/journal.pntd.0005842. eCollection 2017 Oct. No abstract available. PMID 28981505
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Keane E, Funk AL, Shimakawa Y. Systematic review with meta-analysis: the risk of mother-to-child transmission of hepatitis B virus infection in sub-Saharan Africa. Aliment Pharmacol Ther. 2016 Nov;44(10):1005-1017. doi: 10.1111/apt.13795. Epub 2016 Sep 15. PMID 27630001
- [Background] Edmunds WJ, Medley GF, Nokes DJ, O'Callaghan CJ, Whittle HC, Hall AJ. Epidemiological patterns of hepatitis B virus (HBV) in highly endemic areas. Epidemiol Infect. 1996 Oct;117(2):313-25. doi: 10.1017/s0950268800001497. PMID 8870629
- [Background] Breakwell L, Tevi-Benissan C, Childs L, Mihigo R, Tohme R. The status of hepatitis B control in the African region. Pan Afr Med J. 2017 Jun 22;27(Suppl 3):17. doi: 10.11604/pamj.supp.2017.27.3.11981. eCollection 2017. PMID 29296152
- [Background] Wilson P, Parr JB, Jhaveri R, Meshnick SR. Call to Action: Prevention of Mother-to-Child Transmission of Hepatitis B in Africa. J Infect Dis. 2018 Mar 28;217(8):1180-1183. doi: 10.1093/infdis/jiy028. PMID 29351639
- [Background] Andersson MI, Rajbhandari R, Kew MC, Vento S, Preiser W, Hoepelman AI, Theron G, Cotton M, Cohn J, Glebe D, Lesi O, Thursz M, Peters M, Chung R, Wiysonge C. Mother-to-child transmission of hepatitis B virus in sub-Saharan Africa: time to act. Lancet Glob Health. 2015 Jul;3(7):e358-9. doi: 10.1016/S2214-109X(15)00056-X. No abstract available. PMID 26087980
- [Background] Klingler C, Thoumi AI, Mrithinjayam VS. Cost-effectiveness analysis of an additional birth dose of Hepatitis B vaccine to prevent perinatal transmission in a medical setting in Mozambique. Vaccine. 2012 Dec 17;31(1):252-9. doi: 10.1016/j.vaccine.2012.08.007. Epub 2012 Aug 15. PMID 22902676
- [Background] Poovorawan Y, Sanpavat S, Pongpunlert W, Chumdermpadetsuk S, Sentrakul P, Safary A. Protective efficacy of a recombinant DNA hepatitis B vaccine in neonates of HBe antigen-positive mothers. JAMA. 1989 Jun 9;261(22):3278-81. PMID 2523981
- [Background] Wong VC, Ip HM, Reesink HW, Lelie PN, Reerink-Brongers EE, Yeung CY, Ma HK. Prevention of the HBsAg carrier state in newborn infants of mothers who are chronic carriers of HBsAg and HBeAg by administration of hepatitis-B vaccine and hepatitis-B immunoglobulin. Double-blind randomised placebo-controlled study. Lancet. 1984 Apr 28;1(8383):921-6. doi: 10.1016/s0140-6736(84)92388-2. PMID 6143868
- [Background] Tsega E, Tafesse B, Nordenfelt E, Wolde-Hawariat G, Hansson BG, Lindberg J. Immunogenicity of hepatitis B vaccine simultaneously administered with the expanded programme on immunisation (EPI). J Med Virol. 1990 Dec;32(4):232-5. doi: 10.1002/jmv.1890320407. PMID 2150529
- [Background] Apiung T, Ndanu TA, Mingle JA, Sagoe KW. Hepatitis B virus surface antigen and antibody markers in children at a major paediatric hospital after the pentavalent DTP-HBV-Hib vaccination. Ghana Med J. 2017 Mar;51(1):13-19. doi: 10.4314/gmj.v51i1.3. PMID 28959067
- [Background] Abu-Raya B, Kollmann TR, Marchant A, MacGillivray DM. The Immune System of HIV-Exposed Uninfected Infants. Front Immunol. 2016 Sep 28;7:383. doi: 10.3389/fimmu.2016.00383. eCollection 2016. PMID 27733852
- [Background] Njom Nlend AE, Nguwoh PS, Ngounouh CT, Tchidjou HK, Pieme CA, Otele JM, Penlap V, Colizzi V, Moyou RS, Fokam J. HIV-Infected or -Exposed Children Exhibit Lower Immunogenicity to Hepatitis B Vaccine in Yaounde, Cameroon: An Appeal for Revised Policies in Tropical Settings? PLoS One. 2016 Sep 22;11(9):e0161714. doi: 10.1371/journal.pone.0161714. eCollection 2016. PMID 27656883
- [Derived] Tulenko SE, Ngimbi P, Mwandagalirwa K, Tabala M, Matondo J, Ntambua S, Mbonze N, Mbendi C, Luhata C, Jhaveri R, Edwards JK, Becker-Dreps S, Moormann AM, Kaba D, Yotebieng M, Parr JB, Gower EW, Thompson P. Immunogenicity of a Birth Dose of Hepatitis B Vaccine in Kinshasa, Democratic Republic of Congo: A Randomised, Controlled Trial. J Viral Hepat. 2024 Dec;31(12):795-807. doi: 10.1111/jvh.14003. Epub 2024 Sep 24. PMID 39314125
- See also: World Health Organization Global Hepatitis Report, 2017 — https://www.who.int/hepatitis/publications/global-hepatitis-report2017/en/
- See also: Congo Democratic Republic: Demographic and Health Survey, 2013-2014 - Final Report — https://dhsprogram.com/publications/publication-FR300-DHS-Final-Reports.cfm